CLINICAL TRIAL: NCT03245827
Title: Hypogonadotropic Hypogonadism in Obese Young Males
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: not enough recruitment
Sponsor: Sandeep Singh Dhindsa, M.D., F.A.C.E (Other)
Responsible Party: Sponsor-Investigator, Sandeep Singh Dhindsa, M.D., F.A.C.E, Professor, St. Louis University
Organization: St. Louis University (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 28389
Record Dates: First submitted 2017-08-03; First posted 2017-08-10 (Actual); Results first posted 2022-06-29 (Actual); Last update posted 2022-06-29 (Actual); Status verified 2022-06

CONDITIONS: Hypogonadism, Hypogonadotropic
MeSH Terms: conditions — Hypogonadism | interventions — Clomiphene; Exercise

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (4):
- Obese males with hypogonadism-active (Active Comparator): Subjects will be randomized to receive clomiphene capsules
  Interventions: Drug: Clomiphene
- Obese males with hypogonadism-placebo (Placebo Comparator): Subjects will be randomized to receive placebo capsules
  Interventions: Drug: Placebo
- Obese males with normal testosterone (No Intervention): comparison group
- lean males with normal testosterone (No Intervention): comparison group

INTERVENTIONS:
Drug: Clomiphene — clomiphene capsule 25mg twice a week
  Other Names: active
  Arms: Obese males with hypogonadism-active
Drug: Placebo — placebo capsule 25mg twice a week
  Arms: Obese males with hypogonadism-placebo

SUMMARY:
Obesity can lead to low testosterone concentrations in young men. This study will study the effects of low testosterone in those men and the result of treating them with clomiphene.

DETAILED DESCRIPTION:
The prevalence of obesity has increased in children over the past few decades. Approximately 20% of adolescent boys are now considered obese. It is well accepted that obese children are at increased risk for high blood pressure, lipid abnormalities and type 2 diabetes. Recent studies have uncovered yet another undesirable effect of obesity. The testosterone levels of obese boys are only half those of lean boys at completion of puberty. Testosterone is important for muscle and bone development. Men with low testosterone are at higher risk of insulin resistance and inflammation, which lead to type 2 diabetes and heart disease. Since testosterone is the major reproductive hormone, these obese boys are at risk of decreased fertility. Men are supposed to achieve their peak testosterone levels at puberty. Thereafter, there is a decline in testosterone levels at the rate of 2% per year for the rest of life. Thus there is a clear need to develop a deeper understanding of low testosterone in these males who are entering their peak fertility years. There are no approved treatments for this disorder. The investigators propose to conduct a randomized placebo controlled trial to evaluate the effect of treatment with clomiphene in obese young men(age 18-30 years) who have low testosterone concentrations. Clomiphene is a drug that increases testosterone concentrations and possibly increases sperm production. In contrast, testosterone replacement therapy decreased fertility and cannot be used in young men. Investigators will study the effect of treatment with clomiphene or placebo tablets for 12 weeks in 30 subjects. The study will evaluate:-

1. testicular function: Testosterone and two proteins secreted by testis(insulin like factor 3 and inhibin B) will be measured in the blood before and after treatment with clomiphene or placebo.
2. insulin resistance: Investigators will measure insulin and glucose levels in the blood.
3. inflammation: Investigators will measure proteins that induce inflammation.

ELIGIBILITY:
Inclusion Criteria:

* Males
* Age 18-30 years inclusive will be recruited.

A total of 90 males will be recruited:-

* 30 obese males (defined as BMI ≥30 kg/m2) with HH,
* 30 obese males with normal FT concentrations and
* 30 lean males (defined as BMI <25 kg/m2) with normal FT concentrations.

Exclusion Criteria:

* Use of androgens, clomiphene, hCG, aromatase inhibitors or over the counter health supplements which contain androgens currently or in the past 6 months
* Hematocrit > 50%
* Congestive heart failure
* currently suffering from depression
* type 1 diabetes
* Hepatic disease (transaminase > 3 times normal) or cirrhosis
* Renal impairment (eGFR<30 ml/min/1.73m2)
* HIV or Hepatitis C positive status
* Participation in any other concurrent clinical trial
* currently suffering from foot ulcer, significant periodontal disease or any other chronic infectious condition

Ages: 18 Years to 30 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — males
Enrollment: 9 (Actual)
Dates: Start 2019-04-01 (Actual); Primary Completion 2021-10-29 (Actual); Study Completion 2021-10-29 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: sandeep dhindsa, md, Principal Investigator — St. Louis University
Locations (1):
- Saint Louis Univeristy, St Louis, Missouri, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Obese Males With Hypogonadism-active | Obese Males With Hypogonadism-placebo | Obese Males With Normal Testosterone | Lean Males With Normal Testosterone
Started | 1 | 0 | 3 | 5
Completed | 1 | 0 | 3 | 5
Not Completed | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: no subjects were recruited in placebo group
Groups:
- Total: Total of all reporting groups
Arm/Group | Obese Males With Hypogonadism-active | Obese Males With Hypogonadism-placebo | Obese Males With Normal Testosterone | Lean Males With Normal Testosterone | Total
Number analyzed (Participants) | 1 | 0 | 3 | 5 | 9
Age, Continuous [Mean (Standard Deviation); unit: years] | 22 (0) |  | 28 (2) | 21.8 (1.8) | 23.9 (3.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0 | 0 | 0
  Male | 1 | 0 | 3 | 5 | 9
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 2 | 2
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 0 | 0
  White | 1 | 0 | 3 | 3 | 7
  More than one race | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Serum Free Testosterone
Description: after clomiphene or placebo treatment
Time Frame: 12 weeks
Population: Only one volunteer was randomized.
Measure: Mean (Standard Deviation); unit: pg/ml
Arm/Group | Obese Males With Hypogonadism-active | Obese Males With Hypogonadism-placebo
Number analyzed (Participants) | 1 | 0
pg/ml | 85 (NA) — NA is used for standard deviation because there was only one volunteer. |

ADVERSE EVENTS:
Time Frame: 3 months
Description: no subjects were recruited in placebo group
Arm/Group | Obese Males With Hypogonadism-active | Obese Males With Hypogonadism-placebo | Obese Males With Normal Testosterone | Lean Males With Normal Testosterone
All-Cause Mortality (participants affected / at risk) | 0/1 | 0/0 | 0/3 | 0/5
Serious Adverse Events (participants affected / at risk) | 0/1 | 0/0 | 0/3 | 0/5
Other Adverse Events (participants affected / at risk) | 0/1 | 0/0 | 0/3 | 0/5

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-06-02): https://cdn.clinicaltrials.gov/large-docs/27/NCT03245827/Prot_SAP_001.pdf